CLINICAL TRIAL: NCT06861348
Title: Effectiveness and Safety of Inotuzumab Ozogamicin±Donor Lymphocyte Infusion for Relapsed B Cell Acute Lymphoblastic Leukemia/Lymphoblastic Lymphoma After Allogeneic Hematopoietic Stem Cell Transplantation：Phrase II, Multicenter Study
Brief Title: Effectiveness and Safety of InO±DLI for Relapsed B-ALL/LBL After Allo-HSCT
Acronym: ZJU-HSCT-INO
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Principal Investigator, Yi Luo, Clinical Professor, First Affiliated Hospital of Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT20240086C-X1
Record Dates: First submitted 2025-03-03; First posted 2025-03-06 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2024-12

CONDITIONS: Leukemia, Lymphocytic, Acute
Keywords: Inotuzumab Ozogamicin; Donor Lymphocyte Infusion; Relapsed B cell Acute Lymphoblastic Leukemia; Allogeneic Hematopoietic Stem Cell Transplantation
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Burkitt Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Ino±DLI regimen (Experimental): 1. InO induction：the first cycle: 0.8mg/m2, intravenous infusion, d1; 0.5 mg/m2, intravenous infusion, d8, d15. 2.InO consolidation：If CR/CRi was reached after induction, the second cycle :0.5mg/m2, intravenous infusion, d1, d8, d15; If CR/CRi is not reached, Cycle 2 :0.8mg/m2, IV infusion, d1; 0.5 mg/m2, intravenous infusion, d8, d15. 3. DLI: CD3 positive cells 1x10^7/kg; DLI indication: no previous grade III-IV aGVHD, negative HLALOSS test and no present aGVHD and cGVHD.
  Interventions: Drug: Inotuzumab Ozogamicin±Donor Lymphocyte Infusion

INTERVENTIONS:
Drug: Inotuzumab Ozogamicin±Donor Lymphocyte Infusion — Participants will receive Ino±DLI regimen:
  * ① InO induction dose: the first cycle: 0.8mg/m2, intravenous infusion, d1; 0.5 mg/m2, intravenous infusion, d8, d15;
  * ② If CR/CRi was reached after induction, the second cycle :0.5mg/m2, intravenous infusion, d1, d8，d15; If CR/CRi is not reached, Cycle 2 :0.8mg/m2, IV infusion, d1; 0.5 mg/m2, intravenous infusion, d8, d15;
  * ③DLI dose: CD3 positive cells 1x10^7/kg; DLI indication: no previous grade III-IV aGVHD, negative HLALOSS test and no present aGVHD and cGVHD;
  * Lumbar puncture: cytarabine 50mg+dexamethasone 5mg+methotrexate 10mg, intrathecal injection, once a month after remission, a total of 4-6 courses of treatment.

SUMMARY:
B cell acute lymphoblastic leukemia (B-ALL)/Lymphoblastic lymphoma (LBL) is a hematological malignancy caused by malignant transformation and clonal expansion of B-lineage precursor cells. Allogeneic hematopoietic stem cell transplantation (allo-HSCT) remains a potential curable therapy for ALL, especially for high-risk ALL patients. However, post-HSCT recurrence is the primary cause of transplant failure and salvage treatment option for this patient population are very limited. Current data showed that the CR rate and overall survival (OS) in adults with ALL who relapse after transplantation are as low as 30% and 25%, respectively, and the prognosis is extremely dismal. Some researchers have successfully salvage treated relapsed B-ALL patients after transplantation with donor lymphocyte infusions (DLI), but the response rate of DLI alone is usually less than 10%, with increased risk of Graft-Versus-Host Disease (GvHD). In the immunotherapy era, the introduction of immuno-designed therapies like bispecific antibody constructs, antibody conjugates, as well as chimeric antigen receptor T cell (CAR-T) therapy, have immensely broadened the treatment landscape of relapsed or refractory (r/r) B-ALL. Inotuzumab ozogamicin (InO) is a CD22-targeted monoclonal antibody conjugated to the cytotoxic antibiotic calicheamicin. Based on the pivotal Phase III INO-VATE clinical trial published in N Engl J Med in 2016, compared to standard chemotherapy, 73% (64/88) of r/r B-ALL patients treated with InO achieved CR/CRi in the first cycle. Superior CR duration, OS and relapse free survival (RFS) was also observed in the InO group. Subgroup analysis showed that the treatment benefits were consistent for patients who relapsed after allo-HSCT. Moreover, a single-center retrospective study attempted to salvage treat relapsed B-ALL patients after transplantation with combined InO and DLI, results showed that six out of eight patients achieved CR after the first InO course and 75% of patients obtained MRD negativity after the second course, which is quite satisfactory. Therefore, we designed a Phase II clinical study of InO combined with or without DLI in patients with recurrent acute B-ALL/LBL after allo-HSCT, with expectation to increase CR rate and improve long-term survival.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 14-65 years, male or female;
2. Participants with CD22 positive B-ALL/LBL who relapsed after allo-HSCT from a related or unrelated donor (regardless of CD22 expression);
3. ECOG physical status score 0~3, Karnofsky score ≥70;
4. No active grade III/IV graft-versus-host disease (GvHD) or any active liver GvHD, no history of venous occlusive disease (VOD); No active GvHD and no previous history of VOD;
5. Creatinine clearance rate≥50 mL/min (estimate by Cockcroft-Gault Equation);
6. Liver function: alanine transaminase (ALT) and aspartate aminotransferase (AST)≤ 3×upper limit of normal (ULN), and total bilirubin ≤ 2×ULN;
7. Left ventricular ejection fraction (LVEF) ≥50% as measured by echocardiography;
8. Estimated life expectancy >3 months;
9. Participants voluntarily participate in clinical trial; Understand and know this study, sign an informed consent form, and be willing to follow all experimental procedures.

Exclusion Criteria:

1. Allergic or with a history of serious adverse reactions to drugs or drugs with similar chemical structure in this study;
2. Women who are pregnant or breastfeeding, as well as those who are unwilling to take effective contraceptive measures;
3. Severe cardiac dysfunction: left ventricular ejection fraction (LVEF) <60%; Or severe arrhythmia: a history of a clinically significant corrected interval (QTc) prolongation (male >450ms; female>470 ms), ventricular tachycardia, atrial fibrillation, second degree atrioventricular block; myocardial infarction and coronary heart disease with clinical symptoms requiring medical treatment within one year before enrollment;
4. Severe pulmonary disorders (obstructive or restrictive ventilation disorder);
5. Severe liver function impairment: ALT, AST, or TBIL is more than 3 times higher than the upper limit of normal value (ULN);
6. Severe renal impairment: serum Cr is more than 2 times higher than the upper limit of normal (ULN); Or 24-hour urinary creatinine clearance <50ml/min;
7. Participants with active infection or active bleeding who were deemed intolerance to InO treatment by the investigators;
8. A history of new thrombosis, embolism, cerebral hemorrhage or other diseases within one year before enrollment;
9. Participants suffer from known or other mental disorders that investigators are unable to obtain informed consent and may interfere with their ability to comply with research requirements;
10. A history of major organ surgery within the past six weeks;
11. Drug abuse or chronic alcohol abuse that may affect the study results;
12. Participants with a history of organ transplantation other than HSCT (except BMT);
13. Other situations identified by the investigator as unsuitable to participate in the study.

Ages: 14 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 23 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
complete remission rate (CRR) | 1 month after InO treatment
  CR was defined as bone marrow (BM) lymphoblasts≤5%, no evidence of active disease, and complete recovery of peripheral blood counts (platelet count >100×109/L, absolute neutrophil count >1×109/L); CRi was defined as BM lymphoblasts ≤5%, no evidence of active disease, and incomplete recovery of peripheral blood counts (platelet count>50×109/L and absolute neutrophil count >0.5×109/L). CR rate after InO treatment will be recorded.

SECONDARY OUTCOMES:
Duration of remission (DOR) | 2 year
  The period from the first evaluation of CR to the first evaluation of PD or death of any cause.
Overall survival (OS) | 2 years
  The period from the first infusion to any cause of death.
Progression-free survival (PFS) | 2 years
  The period from the day when the participant receives Ino treatment to the first recorded disease progression (whether treated or not) or death of any cause, which occurs first.
Cumulative incidence of disease relapse or progression | 2 year
  All patients will be tracked from Day 0 to date of first objective disease progression, death from any cause, or last patient evaluation. Patients who have not progressed or died will be censored at the last date they were assessed and deemed free of relapse or progression.
Cumulative incidence of transplant-related nonrelapse mortality (NRM) | 2 year
  All patients will be tracked from Day 0 to date of first objective disease progression, death from any cause, or last patient evaluation. Patients who have not progressed or died will be censored at the last date they were assessed and deemed free of relapse or progression.
Incidence of Treatment Related adverse events (AEs) | 2 year
  Incidence of Treatment Related AEs, AEs of special interest and serious adverse events (SAEs) assessed by NCI-CTCAE v5.0 criteria.

OTHER OUTCOMES:
Clonal evolution | 6 month
  Using a single-cell DNA sequencing to report the clonal architecture and mutational histories before and after InO treatment.
Levels of bone marrow B lymphocyte subsets | 6 month
  Percentage of diverse B-cell subsets in bone marrow will be detected by FCM after Ino treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Yi Luo, M.D., Principal Investigator — First Affilaated Hospital of Medical School of Zhejiang University
Locations (1):
- The First Affiliated Hospital, College of Medicine, Zhejiang University, Hangzhou, China

IPD SHARING:
Plan to Share IPD: No